CLINICAL TRIAL: NCT04785638
Title: An Open-label Safety and Pharmacokinetic Study of INL-001 in Adults Following Open Ventral Hernia Repair, Abdominoplasty, Open Abdominal Hysterectomy, Laparoscopic-assisted Colectomy, and Reduction Mammoplasty
Brief Title: An Open-label Safety and Pharmacokinetic Study of INL-001 in Adults Following Various Open Soft-Tissue Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innocoll (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN-CB-025
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative; Hernia, Ventral; Abdominoplasty; Hysterectomy; Colectomy; Reduction Mammoplasty
Keywords: Pain; Analgesia; Postoperative; Hernia; Abdominoplasty; Tummy tuck; Hysterectomy; Colectomy; Bupivacaine; Postsurgical; Implant; Safety; Efficacy; Pharmacokinetic; Opioid; Nonopioid; Post-operative; Post-surgical; Surgery; Soft tissue; Open-label; Phase 3; Local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Hernia, Ventral; Pain; Agnosia; Hernia | interventions — Bupivacaine; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INL-001 (bupivacaine hydrochloride) implant (Experimental): INL-001 (bupivacaine hydrochloride) implant
  Interventions: Combination Product: INL-001 (bupivacaine hydrochloride) implant

INTERVENTIONS:
Combination Product: INL-001 (bupivacaine hydrochloride) implant — INL-001 (bupivacaine hydrochloride) implant
  Other Names: XARACOLL (bupivacaine hydrochloride) Implant

SUMMARY:
This is a multicenter, Phase 3, open-label, safety, tolerability, and characterization of pharmacokinetics study of the INL 001 (bupivacaine HCl) implant, at 300 mg, in patients following various soft-tissue surgeries: open ventral hernia repair, abdominoplasty, open abdominal hysterectomy, laparoscopic-assisted colectomy, and reduction mammoplasty.

DETAILED DESCRIPTION:
This is a multicenter, Phase 3, open-label, safety, tolerability, and characterization of pharmacokinetics study of the INL-001 (bupivacaine HCl) implant, at 300 mg, in patients following various soft-tissue surgeries: open ventral hernia repair, abdominoplasty, open abdominal hysterectomy, laparoscopic-assisted colectomy, and reduction mammoplasty. After a screening period, eligible patients will undergo study surgery under general anesthesia and have INL-001 implanted intraoperatively. Efficacy is also an exploratory measure in this study.

The study includes a screening period, an inpatient period (preoperative, intraoperative, postoperative) of approximately 5 days, and an outpatient follow-up period (up to 30 days after treatment). Posttreatment safety and/or efficacy assessments will be made throughout the study and as specifically scheduled through 96 hours posttreatment, on day 7 (telephone), on day 15 (clinic visit), and on day 30 (clinic visit). Unless the investigator determines further hospitalization is necessary, patients will be discharged approximately 96 hours posttreatment (inpatient day 5).

During the screening period, all patients will undergo eligibility and other screening and safety assessments. In addition, the investigator will administer the Pain Catastrophizing Scale (screening only) as an exploratory measure and the 15-item Quality of Recovery (QoR-15) questionnaire (baseline).

Adverse event and concomitant medication information, including use of rescue pain medication, will be collected throughout the study (inpatient and outpatient). Surgical wound healing/grading assessments and assessment for signs and symptoms potentially indicative of systemic bupivacaine toxicity will be made.

Blood samples for pharmacokinetic assessments will be collected from patients at multiple time points for the measurement of concentrations of bupivacaine in plasma.

After surgery, patient reports of pain intensity using an 11-point numeric pain rating scale (NPRS) will be recorded at multiple time points through 96 hours posttreatment. Patients will be permitted rescue medication (oral and/or intravenous) to manage breakthrough pain when it occurs. The QoR-15 questionnaire and Patient Global Assessment (for pain control) will be administered on an inpatient basis and on day 7. The Opioid Related Symptom Distress Scale will be administered on an inpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index of 18-35 kg/m2.
* Has a planned (nonemergency) open ventral hernia repair, abdominoplasty (with rectus sheath plication, in the opinion of the surgeon), open abdominal hysterectomy, laparoscopic-assisted colectomy, or reduction mammoplasty to be conducted using standard surgical technique under general anesthesia.
* Has the ability and willingness to comply with all study procedures including being domiciled for at least 96 hours after surgery.
* Is willing to use opioid analgesia, if needed.

Exclusion Criteria:

* Has a known hypersensitivity to amide-type local anesthetics, fentanyl, morphine, oxycodone, acetaminophen, NSAIDs, or bovine products.
* Is scheduled for other significant concurrent surgical procedures (eg, cholecystectomy or additional cosmetic procedures concurrent with abdominoplasty).
* Has used an opioid analgesic on an extended daily basis (≥5 mg oral morphine equivalents per day for 3 or more days a week) within 4 weeks before surgery and/or chronically uses pain medication.
* Has any chronic painful condition (eg, fibromyalgia), as determined by the investigator, that may confound the assessment of pain associated with the study surgery.
* For open hernia repair, has open ventral hernia with primary suture repair and mesh placement requiring an incisional length greater than 12 cm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability | Day 1 through Day 30
  The primary objective of the study is to evaluate the safety and tolerability of the INL-001 implant in patients. Measured by frequency and incidents of adverse events.

SECONDARY OUTCOMES:
Cmax | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  Maximum (peak) plasma concentration
Tmax | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  Time to maximum (peak) plasma concentration
Tlag | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  Lag-time
t½ Terminal Half life | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  Terminal Half life
λz | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  Terminal phase rate constant
AUC | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  Area under the plasma concentration-time curve from Time 0 to last time of last quantifiable plasma concentration (AUC0-last)
AUC0-∞ | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48, 72 and 96 hours
  AUC from Time 0 to infinity

OTHER OUTCOMES:
SPI24 | 0 to 24 hours
  Time-weighted sum of pain intensity from Time 0 through 24 hours (SPI24). Lower score has a better outcome. Pain Intensity was assessed by the subject using the 11-point NRS, where 0 indicated "no pain" and 10 indicated "worst pain possible". Minimum value would be "0" and Maximum value would be 240. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI24 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
SPI48 | 0 to 48 hours
  Time-weighted sum of pain intensity from Time 0 through 48 hours (SPI48). Lower score has a better outcome. Pain Intensity was assessed by the subject using the 11-point NRS, where 0 indicated "no pain" and 10 indicated "worst pain possible". Minimum value would be "0" and Maximum value would be 480. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI48 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
SPI72 | 0 to 72 Hours
  Time-weighted sum of pain intensity from Time 0 through 72 hours (SPI72) A lower score is a better outcome. Pain Intensity was assessed by the subject using the 11-point NRS, where 0 indicated "no pain" and 10 indicated "worst pain possible" Minimum value would be "0" and Maximum value would be 720. Time-weighted SPI is calculated as the sum of the pain intensities between successive time points (i.e., if SPI72 = ∑[PI x (time t - time t-1)], where "t" represents a given time point,"t-1" represents the previous time point, and time is expressed in hours). This represents the AUC (Area Under the Curve) of the pain intensities when calculated with the trapezoidal rule.
Total use of opioid rescue analgesia | 0 to 24 hours postoperatively
  Total use of opioid rescue analgesia (mg equivalent) -higher score means more analgesia was needed and worse outcome
Total use of opioid rescue analgesia | 0 to 72 hours postoperatively
  Total use of opioid rescue analgesia (mg equivalent) -higher score means more analgesia was needed and worse outcome
Total use of opioid rescue analgesia | 0 to 48 hours postoperatively
  Total use of opioid rescue analgesia (mg equivalent) -higher score means more analgesia was needed and worse outcome
Time to discharge from the postanesthesia care unit (PACU) | Immediately after the intervention/procedure/surgery
  Time to discharge from the PACU
Opioid-related Symptom Distress Scale (OR-SDS) | 24, 48, 72, and 96 hours posttreatment
  The OR-SDS is a measurement tool to assess patient experience following opioid use in the postoperative setting.
15-item Quality of Recovery (QoR-15) Questionnaire | 24, 48, 72, and 96 hours, and day 7 posttreatment
  The 15-item Quality of Recovery (QoR-15) Questionnaire s a surgical recovery assessment tool. The QoR-15 assesses postsurgical recovery from the patient's perspective and incorporates all 5 dimensions of health patient support, comfort, emotions, physical independence, and pain. Investigator judgement will be used to determine if a positive finding on the QoR-15 is clinically significant and reportable as an adverse event.
Patient Global Assessment (PGA) as Related to Postoperative Pain | 24, 48, 72, and 96 hours, and day 7 posttreatment
  The PGA will be administered by study staff who ask patients to rate "how well your pain has been controlled during the study" on a 5 point nominal scale: 0-poor, 1-fair, 2-good, 3-ery good, or 4-excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Arriaga, Study Director — Lotus Clinical Research
Locations (8):
- United States (8):
  - North Alabama Medical Center, Florence, Alabama
  - Helen Keller Hospital, Sheffield, Alabama
  - Lotus Clinical Research, Pasadena, California
  - Midwest Clinical Research, Dayton, Ohio
  - Daneshvari Solanki, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Memorial Hermann, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No